CLINICAL TRIAL: NCT00615589
Title: Allogeneic Hematopoietic Stem Cell Transplantation For The Treatment Of High Risk Multiple Myeloma With Reduced Toxicity Myeloablative Conditioning Regimen
Brief Title: Stem Cell Transplantation To Treat High Risk Multiple Myeloma With Reduced Toxicity Myeloablative Conditioning Regimen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: umcc 2007.074; HUM00014029
Record Dates: First submitted 2008-01-22; First posted 2008-02-14 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia
Keywords: Stage II/III Multiple Myeloma(within 10 months from diagnosis); high risk; relapse; persistent
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Recurrence | interventions — fludarabine; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flu-Bu4 (Experimental): Fludarabine Busulfan chemotherapy regimen(Flu-Bu4), followed by allogeneic stem cell transplant from best available, matched donor.
  Interventions: Drug: Fludarabine/Busulfan x 4 days; Procedure: stem cell transplant

INTERVENTIONS:
Drug: Fludarabine/Busulfan x 4 days — * Fludarabine: 40 mg/m2/day in NS, administered IV over 30 minutes on days -5, -4, -3, and -2 pre-transplant.
  * Busulfan: 3.2 mg/kg IV daily in NS over 4 hours on days -5, -4, -3, and -2.
  The Fludarabine shall be administered prior to the Busulfan each day.
Procedure: stem cell transplant — Allogeneic, peripheral blood stem cell transplant

SUMMARY:
Standard therapy for multiple myeloma (MM) usually includes an autologous bone marrow stem cell transplant - a procedure where the patient is treated with high dose chemotherapy and then their own (autologous) stem cells are transplanted back into their body. Patients with multiple myeloma and high risk genes, always relapse after an autologous transplant and often die within two years from the time of their transplant. A different type of transplant allogeneic) using donor cells, may work better for high-risk Multiple Myeloma, because the donor cells may help kill the lymphoid cancer cells.

This study will investigate if a matched donor stem cell transplant using a newer, reduced toxicity, chemotherapy (Flu-Bu4) is a feasible option for patients with high risk, Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Biologic high risk Multiple Myeloma:

  * Stage II/III Multiple Myeloma, any of: t(4; 14), t(14; 16),(14:20) by Fish; 17P- by conventional cytogenetics or Fish; ∆13 by conventional cytogenetics; Hypodiploidy by conventional cytogenetics.

    * Relapsed or persistent multiple myeloma after ASCT.
    * Persistent multiple myeloma, regardless of previous therapies.
    * Plasma cell leukemia, regardless of previous therapies.
* Age up to 70 years old (less than 71 years old at the date of transplant admission).
* Disease status: in CR, nCR, VGPR, PR or stable disease within 1 month of admission
* Patients with non-secretory and oligosecretory disease are eligible if they meet certain criteria within 2 weeks prior to the transplant.
* Specific renal, liver, cardiac, and pulmonary function requirements(all must be met within 30 days of transplant admission)

Exclusion Criteria:

* Persistent invasive infections, not controlled by antimicrobials.
* HIV-1/HIV-2 or HTLV-1/HTLV-2 seropositivity.
* Uncontrolled medical or psychiatric disorder.
* No response or progressive disease at the time of transplantation.
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Attaphol Pawarode, MD, Principal Investigator — University of Michigan Dept. of Internal Medicine
Locations (1):
- University of Michigan,Department of Internal Med. Hematology- Oncology, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Flu-Bu4: Fludarabine Busulfan chemotherapy regimen (Flu-Bu4), followed by allogeneic stem cell transplant from best available, matched donor.
  Fludarabine/Busulfan x 4 days:
  Fludarabine: 40 mg/m2/day, administered IV over 30 minutes on days -5, -4, -3, and -2 pre-transplant.
  Busulfan: 3.2 mg/kg IV daily over 4 hours on days -5, -4, -3, and -2.
  The Fludarabine shall be administered prior to the Busulfan each day.
Period: Overall Study
Arm/Group | Flu-Bu4
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Flu-Bu4: Fludarabine Busulfan chemotherapy regimen(Flu-Bu4), followed by allogeneic stem cell transplant from best available, matched donor.
  Fludarabine/Busulfan x 4 days:
  Fludarabine: 40 mg/m2/day in NS, administered IV over 30 minutes on days -5, -4, -3, and -2 pre-transplant.
  Busulfan: 3.2 mg/kg IV daily in NS over 4 hours on days -5, -4, -3, and -2.
  The Fludarabine shall be administered prior to the Busulfan each day.
Arm/Group | Flu-Bu4
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 54 [45 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Alive 1 Year Post Transplant
Description: The primary objective is overall survival, one year from the time of transplant.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Flu-Bu4
Number analyzed (Participants) | 22
percentage of patients | 61 [43 to 87]

2. Secondary Outcome: The Percentage of Patients Free From Progression at 1 Year
Description: One of the secondary outcomes that will be measured is progression free survival at 1 Year.
  Progressive Disease (PD) is defined as a >25% increase in serum monoclonal paraprotein, a >25% increase in 24-hour urinary light chain excretion, a >25% increase in plasma cells in bone marrow aspirate, an increase in the size or the development of new bone lesions/soft tissue plasmacytomas, or the development of hypercalcemia.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Flu-Bu4
Number analyzed (Participants) | 22
percentage of patients | 40 [23 to 67]

3. Secondary Outcome: Percentage of Patients With Treatment Related Mortality (TRM)
Time Frame: 100 days, one-year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Flu-Bu4
Number analyzed (Participants) | 22
percentage of patients | 9 [2 to 33]

4. Secondary Outcome: Percentage of Patients With Acute and Chronic Graft Versus Host Disease (GVHD)
Description: Incidence of acute (Stage II-IV and Stage III-IV) and chronic GVHD (any stage) were analyzed.
  Acute GVHD Grading:
  Stage II - Skin, 25-50% BSA (Body Surface Area); Liver, 3.1-6mg/dl bilirubin; Gut, 1000-1500ml/day diarrhea Stage III - Skin, generalized erythroderma; Liver, 6.1-15mg/dl bilirubin; Gut, >1500ml/day diarrhea Stage IV - Skin, bullae; Liver, >15mg/dl bilirubin; Gut, pain +/- ileus
Time Frame: 100 days, 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flu-Bu4
Number analyzed (Participants) | 22
percentage of participants
  Grade II-IV Acute GVHD | 48 [29 to 72]
  Grade III-IV Acute GVHD | 23 [10 to 47]
  Chronic GVHD | 55 [34 to 78]

5. Secondary Outcome: Non Relapse Mortality (NRM) at 1 Year and 3 yearsThe Percentage of Deaths Not Attributable to Disease Relapse or Progression
Description: Non relapse mortality, defined as the percentage of deaths not attributable to disease relapse or progression at 1 year and at 3 years.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of deaths
Arm/Group | Flu-Bu4
Number analyzed (Participants) | 22
percentage of deaths
  NRM at 1 Year | 19 [7 to 44]
  NRM at 3 Years | 29 [13 to 55]

ADVERSE EVENTS:
Arm/Group | Flu-Bu4
Serious Adverse Events (participants affected / at risk) | 13/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flu-Bu4 (N=22)
Allergy/Immunology - Other (Immune system disorders) | 1 (1)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 2 (2)
Cardiac General - Other (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Death, disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Hemorrhage, bladder (Vascular disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1)
Infection, blood (Infections and infestations) | 1 (1)
Infection, lung (Infections and infestations) | 1 (1)
Infection, upper airway (Infections and infestations) | 1 (1)
Infection, UTI (Infections and infestations) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
Pain, headache (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flu-Bu4 (N=22)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 8 (9)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2)
Hypertension (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 6 (6)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5)
Fever (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (5)
Weight gain (Metabolism and nutrition disorders) | 2 (2)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 6 (8)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4 (4)
Gastrointestinal - Other (Specify) (Gastrointestinal disorders) | 3 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3)
Incontinence, anal (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 3 (3)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 6 (7)
Hemorrhage, GI (Gastrointestinal disorders) | 3 (3)
Hemorrhage, GI (Gastrointestinal disorders) | 2 (2)
Hemorrhage, GU (Renal and urinary disorders) | 2 (3)
Hemorrhage, GU (Renal and urinary disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infection - Other (Specify) (Infections and infestations) | 5 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 3 (5)
Edema: head and neck (General disorders) | 2 (2)
Edema: limb (General disorders) | 5 (5)
Edema: trunk/genital (General disorders) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 2 (2)
Alkaline phosphatase (Investigations) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Confusion (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 6 (7)
Mood alteration, anxiety (Psychiatric disorders) | 2 (2)
Neurology - Other (Nervous system disorders) | 3 (4)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 7 (7)
Dry eye syndrome (Eye disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 3 (3)
Pain, back (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain, bone (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain, headache (Nervous system disorders) | 5 (6)
Pain, neck (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain, pelvis (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain - Other (General disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bladder spasms (Renal and urinary disorders) | 2 (3)
Renal failure (Renal and urinary disorders) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (2)
Syndromes - Other (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes